CLINICAL TRIAL: NCT06933823
Title: Dietary Modification Intervention Involving Family Support (FamNUTRI) for Managing Sarcopenic Obesity Among Community-dwelling Older Adults: a Pilot Randomized Controlled Trial
Brief Title: Dietary Modification Intervention Involving Family Support (FamNUTRI) for Managing Sarcopenic Obesity Among Community-dwelling Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20241105001
Record Dates: First submitted 2025-04-02; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenic Obesity
Keywords: Sarcopenic Obesity; Dietary intervention; Pilot RCT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded independent assessor will assess the participants' outcomes without knowing their group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FamNUTRI group (Experimental): The experimental FamNUTRI group will receive dietary modification intervention in the older adult centre. A total of 6 face-to-face one-hour bi-weekly sessions of the dietary modification program combined with bi-weekly phone calls for the intervention period of 15 weeks to foster their adherence to the hypocaloric diet with high protein intake will be included in the intervention. They will be asked to invite one of their family members to attend the sessions together.
  Interventions: Behavioral: Dietary modification intervention involving family support
- NUTRI group (Active Comparator): The participants in NUTRI group will receive a total of 6 face-to-face one-hour bi-weekly sessions of the dietary modification program combined with bi-weekly phone calls for the intervention period of 15 weeks to foster their adherence to the hypocaloric diet with high protein intake.
  Interventions: Behavioral: Dietary modification intervention
- Control Group (No Intervention): This control group will not receive any intervention and participants will be instructed to maintain their original dietary habits.

INTERVENTIONS:
Behavioral: Dietary modification intervention involving family support — The intervention includes six one-hour, bi-weekly face-to-face sessions, along with bi-weekly phone calls over 15 weeks, to support participants in adhering to a hypocaloric and high-protein diet. The participants will be asked to invite one of their family members to attend the sessions together. Family members will be engaged in discussions to help enhance the participant's adherence to the recommended diet regimen. The aims of the sessions are to raise awareness among participants and their families about sarcopenia obesity and the recommended dietary modifications, emphasizing the critical role of family in supporting adherence to these changes. It also focuses on boosting participants' motivation, reducing barriers to dietary adjustments, and enhancing family-driven social support to help sustain long-term adherence to the prescribed regimen.
  Arms: FamNUTRI group
Behavioral: Dietary modification intervention — The intervention includes six one-hour, bi-weekly face-to-face sessions, along with bi-weekly phone calls over 15 weeks, to support participants in adhering to a hypocaloric and high-protein diet. The sessions will only focus on educating the participants on following the dietary regimen and addressing the barriers they may encounter during dietary modification without family involving in the intervention.
  Arms: NUTRI group

SUMMARY:
The goal of this pilot RCT is to examine the feasibility and preliminary effects of a dietary modification intervention involving family support (FamNUTRI) on the management of sarcopenic obesity among older people living in the community. The main questions it aims to answer are:

1. Is the intervention feasible and acceptable for community-dwelling older people with sarcopenic obesity?
2. What are the preliminary effects of the intervention on managing sarcopenic obesity in this population?

Researchers will compare the FamNUTRI group, the NUTRI group, and a passive control group to see if the dietary modification intervention with family support has additional benefits over the dietary modification intervention alone and no intervention.

Participants will:

Attend 6 face-to-face one-hour bi-weekly sessions over 15 weeks Receive bi-weekly phone calls to foster adherence to the hypocaloric diet with high protein intake (For the FamNUTRI group) Invite a family member to attend the sessions together

ELIGIBILITY:
Inclusion Criteria:

1. older adults aged 65 years old or above who are living in the community and have not less than 4 shared meals with family weekly
2. having a family member consent to offer support to the study participant
3. diagnosed as having sarcopenic obesity using the diagnostic criteria of Asian Working Group for Sarcopenia (AWGS) for sarcopenia and definition from WHO for obesity for Asian, respectively: 3a)early-stage sarcopenia is defined by meeting one of the following criteria: low handgrip strength <28 kg for men and <18 kg for women, low appendicular skeletal muscle mass (ASM) /height2 < 7 kg/m2 for men and <5.7 kg/m2 for women, or low physical performance with a Short Physical Performance Battery (SPPB) score of < 9; 3b) Obesity is defined by meeting one of the following criteria: BMI ≥25 kg/m2, waist circumference ≥ 90 cm in men and ≥ 80 cm in women, or percentage of body fat >30%
4. ability to read, write and understand Chinese without severe speaking, hearing and vision problems for intervention delivery.

Exclusion Criteria:

1. having any existing disease or condition that affects digestion or food intake, such as severe heart diseases, renal diseases, depression or advanced stages of cancer
2. having medications that impact dietary patterns, digestion, or metabolism
3. following specific dietary pattern or restrictions, such as diabetic diets and renal diets
4. having alcohol addiction defined by Alcohol Use Disorders Identification Test (AUDIT) scoring 8 or above since it may affect their ability and their determination to make changes in dietary modification
5. having medical implants such as a pacemaker since the equipment to carry out bioelectric impedance analysis (Inbody S10) may cause malfunctioning of the implanted devices.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Changes of muscle mass | Change from baseline to the end of intervention at 15 weeks
  Muscle mass (kg) will be measured by using bioelectrical impedance analysis.
Changes of muscle strength | Change from baseline to the end of intervention at 15 weeks
  Handgrip strength (kg) will be measured by using the digital dynamometer.
The Short Physical Performance Battery scale | Change from baseline to the end of intervention at 15 weeks
  The Short Physical Performance Battery (SPPB) measures balance, lower extremity strength and functional capacity. It is a well-established tool for assessing physical function in older adults. It consists of three types of assessments: standing for 10 seconds with feet in three different positions, a 3-meter or 4-meter walking speed test, and the time to rise from a chair for five times. The final total SPPB score ranges from 4 to 12. Scores will be categorized as low performance (4-6), middle performance (7-9) and best performance (10-12).
Change of weight | Change from baseline to the end of intervention at 15 weeks
  Weight will be measured and recorded in kilograms
Height | Change from baseline to the end of intervention at 15 weeks
  Height will be measured and recorded in meters.
Changes of body mass index | Change from baseline to the end of intervention at 15 weeks
  The weight and height will be combined to report BMI in kg/m^2.
Changes of percentage of body fat | Change from baseline to the end of intervention at 15 weeks
  Percentage of body fat will be measured by using bioelectrical impedance analysis.

SECONDARY OUTCOMES:
Mini Nutritional Assessment (MNA) scale | Change from baseline to the end of intervention at 15 weeks
  The Mini Nutritional Assessment (MNA) scale will be used to measure the participants' nutritional status. Scores on the MNA range from 0 to 30, with higher scores indicating better nutritional status. Scoring 24-30 indicates normal nutritional status, scoring 17-23.5 indicates a risk of malnutrition, and scoring less than 17 indicates malnourished.
Dietary Quality International-Index (DQI-I) | Change from baseline to the end of intervention at 15 weeks
  The Dietary Quality International-Index (DQI-I) will be used to measure the dietary quality. The DQI-I assessed four aspects of diet which include variety, adequacy, moderation, and overall balance. Total scores on the DQI-I range from 0 to 100, with higher scores indicating a better quality of diet.
Diet adherence | Change from baseline to the end of intervention at 15 weeks
  Diet adherence will be measured by the protein intake and caloric restriction based on the 3-day dietary record. The adherence to protein intake will be reflected by the protein score in the DQI-I which will be calculated based on participant's 3-day dietary record. Also. the participants' attendance rate in the consultation sessions will be monitored.
Health action process approach(HAPA)Nutrition Self-efficacy Scale | Change from baseline to the end of intervention at 15 weeks
  The Nutrition Self-Efficacy Scale is a component of the Health-Specific Self-Efficacy Scale, created by Ralf Schwarzer and Britta Renner. It consists of 5 items, each rated on a 4-point Likert scale: 1 = Very Uncertain, 2 = Rather Uncertain, 3 = Rather Certain, and 4 = Very Certain. Higher scores indicate greater self-efficacy. The total scores range from 5 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Ying Mak, BSN, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
To maintain confidentiality, all participant information will remain anonymous and replaced with reference codes. The collected data will be securely stored, with physical copies kept in a locked location and electronic files encrypted and accessible only to the research team. All data will be destroyed within seven years following the conclusion of this study.

REFERENCES:
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Zhou X, Perez-Cueto FJA, Santos QD, Monteleone E, Giboreau A, Appleton KM, Bjorner T, Bredie WLP, Hartwell H. A Systematic Review of Behavioural Interventions Promoting Healthy Eating among Older People. Nutrients. 2018 Jan 26;10(2):128. doi: 10.3390/nu10020128. PMID 29373529
- [Background] Gilbert SJ, Zamenopoulos T, Alexiou K, Johnson JH. Involvement of right dorsolateral prefrontal cortex in ill-structured design cognition: an fMRI study. Brain Res. 2010 Feb 2;1312:79-88. doi: 10.1016/j.brainres.2009.11.045. Epub 2009 Nov 27. PMID 19948156
- [Background] Willoughby D, Hewlings S, Kalman D. Body Composition Changes in Weight Loss: Strategies and Supplementation for Maintaining Lean Body Mass, a Brief Review. Nutrients. 2018 Dec 3;10(12):1876. doi: 10.3390/nu10121876. PMID 30513859
- [Background] Villareal DT, Aguirre L, Gurney AB, Waters DL, Sinacore DR, Colombo E, Armamento-Villareal R, Qualls C. Aerobic or Resistance Exercise, or Both, in Dieting Obese Older Adults. N Engl J Med. 2017 May 18;376(20):1943-1955. doi: 10.1056/NEJMoa1616338. PMID 28514618
- [Background] Verjans-Janssen SRB, van de Kolk I, Van Kann DHH, Kremers SPJ, Gerards SMPL. Effectiveness of school-based physical activity and nutrition interventions with direct parental involvement on children's BMI and energy balance-related behaviors - A systematic review. PLoS One. 2018 Sep 27;13(9):e0204560. doi: 10.1371/journal.pone.0204560. eCollection 2018. PMID 30261057
- [Background] Vellas B, Villars H, Abellan G, Soto ME, Rolland Y, Guigoz Y, Morley JE, Chumlea W, Salva A, Rubenstein LZ, Garry P. Overview of the MNA--Its history and challenges. J Nutr Health Aging. 2006 Nov-Dec;10(6):456-63; discussion 463-5. PMID 17183418
- [Background] Trouwborst I, Verreijen A, Memelink R, Massanet P, Boirie Y, Weijs P, Tieland M. Exercise and Nutrition Strategies to Counteract Sarcopenic Obesity. Nutrients. 2018 May 12;10(5):605. doi: 10.3390/nu10050605. PMID 29757230
- [Background] Sammarco R, Marra M, Di Guglielmo ML, Naccarato M, Contaldo F, Poggiogalle E, Donini LM, Pasanisi F. Evaluation of Hypocaloric Diet With Protein Supplementation in Middle-Aged Sarcopenic Obese Women: A Pilot Study. Obes Facts. 2017;10(3):160-167. doi: 10.1159/000468153. Epub 2017 May 20. PMID 28528340
- [Background] Rosland AM, Kieffer E, Israel B, Cofield M, Palmisano G, Sinco B, Spencer M, Heisler M. When is social support important? The association of family support and professional support with specific diabetes self-management behaviors. J Gen Intern Med. 2008 Dec;23(12):1992-9. doi: 10.1007/s11606-008-0814-7. Epub 2008 Oct 15. PMID 18855075
- [Background] Robinson SM, Reginster JY, Rizzoli R, Shaw SC, Kanis JA, Bautmans I, Bischoff-Ferrari H, Bruyere O, Cesari M, Dawson-Hughes B, Fielding RA, Kaufman JM, Landi F, Malafarina V, Rolland Y, van Loon LJ, Vellas B, Visser M, Cooper C; ESCEO working group. Does nutrition play a role in the prevention and management of sarcopenia? Clin Nutr. 2018 Aug;37(4):1121-1132. doi: 10.1016/j.clnu.2017.08.016. Epub 2017 Aug 24. PMID 28927897
- [Background] Peters MDJ, Godfrey C, McInerney P, Khalil H, Larsen P, Marnie C, Pollock D, Tricco AC, Munn Z. Best practice guidance and reporting items for the development of scoping review protocols. JBI Evid Synth. 2022 Apr 1;20(4):953-968. doi: 10.11124/JBIES-21-00242. PMID 35102103
- [Background] Phillips BE, Atherton PJ, Varadhan K, Limb MC, Wilkinson DJ, Sjoberg KA, Smith K, Williams JP. The effects of resistance exercise training on macro- and micro-circulatory responses to feeding and skeletal muscle protein anabolism in older men. J Physiol. 2015 Jun 15;593(12):2721-34. doi: 10.1113/JP270343. Epub 2015 May 14. PMID 25867865
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Nilsson MI, Dobson JP, Greene NP, Wiggs MP, Shimkus KL, Wudeck EV, Davis AR, Laureano ML, Fluckey JD. Abnormal protein turnover and anabolic resistance to exercise in sarcopenic obesity. FASEB J. 2013 Oct;27(10):3905-16. doi: 10.1096/fj.12-224006. Epub 2013 Jun 26. PMID 23804240
- [Background] Muscariello E, Nasti G, Siervo M, Di Maro M, Lapi D, D'Addio G, Colantuoni A. Dietary protein intake in sarcopenic obese older women. Clin Interv Aging. 2016 Feb 5;11:133-40. doi: 10.2147/CIA.S96017. eCollection 2016. PMID 26917955
- [Background] Murton AJ, Marimuthu K, Mallinson JE, Selby AL, Smith K, Rennie MJ, Greenhaff PL. Obesity Appears to Be Associated With Altered Muscle Protein Synthetic and Breakdown Responses to Increased Nutrient Delivery in Older Men, but Not Reduced Muscle Mass or Contractile Function. Diabetes. 2015 Sep;64(9):3160-71. doi: 10.2337/db15-0021. Epub 2015 May 26. PMID 26015550
- [Background] Moser A, Melchior I, Veenstra M, Stoffers E, Derks E, Jie KS. Improving the experience of older people with colorectal and breast cancer in patient-centred cancer care pathways using experience-based co-design. Health Expect. 2021 Apr;24(2):478-490. doi: 10.1111/hex.13189. Epub 2021 Jan 13. PMID 33440059
- [Background] Misra D, Fielding RA, Felson DT, Niu J, Brown C, Nevitt M, Lewis CE, Torner J, Neogi T; MOST study. Risk of Knee Osteoarthritis With Obesity, Sarcopenic Obesity, and Sarcopenia. Arthritis Rheumatol. 2019 Feb;71(2):232-237. doi: 10.1002/art.40692. Epub 2019 Jan 4. PMID 30106249
- [Background] Marshall S, Bauer J, Capra S, Isenring E. Are informal carers and community care workers effective in managing malnutrition in the older adult community? A systematic review of current evidence. J Nutr Health Aging. 2013;17(8):645-51. doi: 10.1007/s12603-013-0341-z. PMID 24097017
- [Background] Marshall S, Agarwal E, Young A, Isenring E. Role of domiciliary and family carers in individualised nutrition support for older adults living in the community. Maturitas. 2017 Apr;98:20-29. doi: 10.1016/j.maturitas.2017.01.004. Epub 2017 Jan 12. PMID 28274324
- [Background] Lo JH, U KP, Yiu T, Ong MT, Lee WY. Sarcopenia: Current treatments and new regenerative therapeutic approaches. J Orthop Translat. 2020 Apr 30;23:38-52. doi: 10.1016/j.jot.2020.04.002. eCollection 2020 Jul. PMID 32489859
- [Background] Liu KSN, Chen JY, Ng MYC, Yeung MHY, Bedford LE, Lam CLK. How Does the Family Influence Adolescent Eating Habits in Terms of Knowledge, Attitudes and Practices? A Global Systematic Review of Qualitative Studies. Nutrients. 2021 Oct 22;13(11):3717. doi: 10.3390/nu13113717. PMID 34835973
- [Background] Lang T, Streeper T, Cawthon P, Baldwin K, Taaffe DR, Harris TB. Sarcopenia: etiology, clinical consequences, intervention, and assessment. Osteoporos Int. 2010 Apr;21(4):543-59. doi: 10.1007/s00198-009-1059-y. Epub 2009 Sep 25. PMID 19779761
- [Background] Lambert CP, Wright NR, Finck BN, Villareal DT. Exercise but not diet-induced weight loss decreases skeletal muscle inflammatory gene expression in frail obese elderly persons. J Appl Physiol (1985). 2008 Aug;105(2):473-8. doi: 10.1152/japplphysiol.00006.2008. Epub 2008 Jun 5. PMID 18535122
- [Background] Kim JE, O'Connor LE, Sands LP, Slebodnik MB, Campbell WW. Effects of dietary protein intake on body composition changes after weight loss in older adults: a systematic review and meta-analysis. Nutr Rev. 2016 Mar;74(3):210-24. doi: 10.1093/nutrit/nuv065. Epub 2016 Feb 16. PMID 26883880
- [Background] Justine M, Azizan A, Hassan V, Salleh Z, Manaf H. Barriers to participation in physical activity and exercise among middle-aged and elderly individuals. Singapore Med J. 2013 Oct;54(10):581-6. doi: 10.11622/smedj.2013203. PMID 24154584
- [Background] Jeloka TK, Dharmatti G, Jamdade T, Pandit M. Are oral protein supplements helpful in the management of malnutrition in dialysis patients? Indian J Nephrol. 2013 Jan;23(1):1-4. doi: 10.4103/0971-4065.107185. PMID 23580797
- [Background] Hatipoglu N, Ozturk A, Mazicioglu MM, Kurtoglu S, Seyhan S, Lokoglu F. Waist circumference percentiles for 7- to 17-year-old Turkish children and adolescents. Eur J Pediatr. 2008 Apr;167(4):383-9. doi: 10.1007/s00431-007-0502-3. Epub 2007 May 9. PMID 17487506
- [Background] Guillet C, Delcourt I, Rance M, Giraudet C, Walrand S, Bedu M, Duche P, Boirie Y. Changes in basal and insulin and amino acid response of whole body and skeletal muscle proteins in obese men. J Clin Endocrinol Metab. 2009 Aug;94(8):3044-50. doi: 10.1210/jc.2008-2216. Epub 2009 May 26. PMID 19470633
- [Background] Goisser S, Kemmler W, Porzel S, Volkert D, Sieber CC, Bollheimer LC, Freiberger E. Sarcopenic obesity and complex interventions with nutrition and exercise in community-dwelling older persons--a narrative review. Clin Interv Aging. 2015 Aug 6;10:1267-82. doi: 10.2147/CIA.S82454. eCollection 2015. PMID 26346071
- [Background] Hill KG, Woodward D, Woelfel T, Hawkins JD, Green S. Planning for Long-Term Follow-Up: Strategies Learned from Longitudinal Studies. Prev Sci. 2016 Oct;17(7):806-18. doi: 10.1007/s11121-015-0610-7. PMID 26453453
- [Background] Heymsfield SB, Gonzalez MC, Shen W, Redman L, Thomas D. Weight loss composition is one-fourth fat-free mass: a critical review and critique of this widely cited rule. Obes Rev. 2014 Apr;15(4):310-21. doi: 10.1111/obr.12143. Epub 2014 Jan 22. PMID 24447775
- [Background] Deutz NE, Bauer JM, Barazzoni R, Biolo G, Boirie Y, Bosy-Westphal A, Cederholm T, Cruz-Jentoft A, Krznaric Z, Nair KS, Singer P, Teta D, Tipton K, Calder PC. Protein intake and exercise for optimal muscle function with aging: recommendations from the ESPEN Expert Group. Clin Nutr. 2014 Dec;33(6):929-36. doi: 10.1016/j.clnu.2014.04.007. Epub 2014 Apr 24. PMID 24814383
- [Background] Ellis KR, Raji D, Olaniran M, Alick C, Nichols D, Allicock M. A systematic scoping review of post-treatment lifestyle interventions for adult cancer survivors and family members. J Cancer Surviv. 2022 Apr;16(2):233-256. doi: 10.1007/s11764-021-01013-x. Epub 2021 Mar 13. PMID 33713302
- [Background] Dondero KR, Falvey JR, Beamer BA, Addison O. Geriatric Vulnerabilities Among Obese Older Adults With and Without Sarcopenia: Findings From a Nationally Representative Cohort Study. J Geriatr Phys Ther. 2022 Jul-Sep 01;46(3):168-173. doi: 10.1519/JPT.0000000000000358. Epub 2022 Aug 18. PMID 35981333
- [Background] Chung JY, Kang HT, Lee DC, Lee HR, Lee YJ. Body composition and its association with cardiometabolic risk factors in the elderly: a focus on sarcopenic obesity. Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):270-8. doi: 10.1016/j.archger.2012.09.007. Epub 2012 Oct 15. PMID 23079031
- [Background] Choi SH, Yang ECL, Tabari S. Solo dining in Chinese restaurants: A mixed-method study in Macao. Int J Hosp Manag. 2020 Sep;90:102628. doi: 10.1016/j.ijhm.2020.102628. Epub 2020 Jul 29. PMID 32834354
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Cava E, Padua E, Campaci D, Bernardi M, Muthanna FMS, Caprio M, Lombardo M. Investigating the Health Implications of Whey Protein Consumption: A Narrative Review of Risks, Adverse Effects, and Associated Health Issues. Healthcare (Basel). 2024 Jan 18;12(2):246. doi: 10.3390/healthcare12020246. PMID 38255133
- [Background] Bevan Jones R, Stallard P, Agha SS, Rice S, Werner-Seidler A, Stasiak K, Kahn J, Simpson SA, Alvarez-Jimenez M, Rice F, Evans R, Merry S. Practitioner review: Co-design of digital mental health technologies with children and young people. J Child Psychol Psychiatry. 2020 Aug;61(8):928-940. doi: 10.1111/jcpp.13258. Epub 2020 Jun 22. PMID 32572961
- [Background] Bethancourt HJ, Rosenberg DE, Beatty T, Arterburn DE. Barriers to and facilitators of physical activity program use among older adults. Clin Med Res. 2014 Sep;12(1-2):10-20. doi: 10.3121/cmr.2013.1171. Epub 2014 Jan 10. PMID 24415748
- [Background] Bauer J, Biolo G, Cederholm T, Cesari M, Cruz-Jentoft AJ, Morley JE, Phillips S, Sieber C, Stehle P, Teta D, Visvanathan R, Volpi E, Boirie Y. Evidence-based recommendations for optimal dietary protein intake in older people: a position paper from the PROT-AGE Study Group. J Am Med Dir Assoc. 2013 Aug;14(8):542-59. doi: 10.1016/j.jamda.2013.05.021. Epub 2013 Jul 16. PMID 23867520
- [Background] Batsis JA, Gill LE, Masutani RK, Adachi-Mejia AM, Blunt HB, Bagley PJ, Lopez-Jimenez F, Bartels SJ. Weight Loss Interventions in Older Adults with Obesity: A Systematic Review of Randomized Controlled Trials Since 2005. J Am Geriatr Soc. 2017 Feb;65(2):257-268. doi: 10.1111/jgs.14514. Epub 2016 Sep 19. PMID 27641543
- [Background] Aryal V, Ghimire D, Kandel S, Majumder A, Manna S. Obesity among Medical Students of a Medical College: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2022 Nov 2;60(255):943-946. doi: 10.31729/jnma.7519. PMID 36705181
- [Background] Anton SD, Manini TM, Milsom VA, Dubyak P, Cesari M, Cheng J, Daniels MJ, Marsiske M, Pahor M, Leeuwenburgh C, Perri MG. Effects of a weight loss plus exercise program on physical function in overweight, older women: a randomized controlled trial. Clin Interv Aging. 2011;6:141-9. doi: 10.2147/CIA.S17001. Epub 2011 Jun 15. PMID 21753869
- [Background] Allen KN, Taylor JS, Kuiper R. Effectiveness of nutrition education on fast food choices in adolescents. J Sch Nurs. 2007 Dec;23(6):337-41. doi: 10.1177/10598405070230060601. PMID 18052519
- See also: Inbody S10 — https://inbodyusa.com/products/inbodys10/
- See also: Food Processor — https://www.trustwell.com/products/food-processor-nutrition-analysis-software/dietitian-purchase/